CLINICAL TRIAL: NCT07325123
Title: An Exploratory Study on the Safety and Efficacy of Malic Acid Supplementation Combined With Immunotherapy in Patients With Solid Tumors
Brief Title: Malic Acid Supplementation Combined With Immunotherapy in Patients With Solid Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chase019
Record Dates: First submitted 2025-09-01; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor Malignancies
MeSH Terms: interventions — malic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dose group (Experimental)
  Interventions: Drug: Malic Acid

INTERVENTIONS:
Drug: Malic Acid — This is a study on the safety and efficacy of malic acid supplementation combined with immunotherapy for anti-tumor treatment in patients with solid tumors. Primary study objective: To determine the oral safety of malic acid. Secondary study objectives: 1. To evaluate the preliminary efficacy of malic acid in the study population. 2. To determine the recommended phase 2 dose (RP2D) of oral malic acid. Exploratory endpoints: Immune indicators including white blood cell count, neutrophil, lymphocyte, monocyte, eosinophil and basophil (count/proportion); metabolic indicators including blood glucose, triglycerides; nutritional indicators including body weight. Starting dose: The proposed starting dose of malic acid (MA) in humans is 30 mg/kg/day (for two immunotherapy cycles). Dose levels: 30 mg/kg/day → 60 mg/kg/day → 90 mg/kg/day (with an incremental increase not exceeding 100%), to be administered after meals.

SUMMARY:
This is a study on the safety and efficacy of malic acid supplementation combined with immunotherapy for anti-tumor treatment in patients with solid tumors. The primary study objective is to determine the oral safety of malic acid; Secondary study objectives: 1. To evaluate the preliminary efficacy of malic acid in the study population. 2. To determine the recommended phase 2 dose (RP2D) of oral malic acid. Exploratory endpoints: Immune indicators including white blood cell count, neutrophil, lymphocyte, monocyte, eosinophil and basophil (count/proportion); metabolic indicators including blood glucose, triglycerides; nutritional indicators including body weight.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years (inclusive), male or female;
* Patients with malignant solid tumors such as colorectal cancer, lung cancer, and melanoma, confirmed by histopathological or cytological examination;
* Patients have at least one measurable lesion;
* Undergoing systematic anti-tumor treatment with immunotherapy;
* Expected survival time ≥ 3 months;
* Basic functions of major organs are norma，laboratory tests meet the following criteria：Hematology (No blood transfusion or blood products administered, and no use of G-CSF or other hematopoietic stimulants for correction within 7 days prior to laboratory testing): Absolute neutrophil count ≥ 1.5×10⁹/L; Platelets ≥ 75×10⁹/L; Hemoglobin ≥ 90g/L. Kidney: Creatinine clearance (CrCl) or estimated glomerular filtration rate (eGFR) > 60ml/min/1.73m² (Cockcroft-Gault formula). Liver: Serum total bilirubin < 1.5×ULN; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5×ULN or ≤ 5×ULN (for subjects with liver metastases); Albumin (ALB) ≥ 30g/L. Coagulation function: International normalized ratio (INR) or prothrombin time (PT) < 1.5×ULN. For subjects receiving anticoagulant therapy, it is acceptable as long as PT is within the intended range for the anticoagulant used.l;
* For female subjects of childbearing age during the screening period, the serum pregnancy test result must be negative; female/male subjects of reproductive potential must be willing to use reliable contraceptive methods throughout the entire study period (i.e., from signing the informed consent form to 90 days after the last administration of the study drug), including but not limited to: abstinence, vasectomy of the male partner, female sterilization, effective intrauterine devices (IUDs), and effective contraceptive medications.
* Patients voluntarily participate in this study, sign the informed consent form, and have good compliance.

Exclusion Criteria:

* Subjects who have not recovered from adverse events caused by any intervention to ≤ Grade 1 (except for alopecia, hearing impairment, and Grade ≤ 2 neurological or endocrine disorders requiring replacement therapy) prior to the first dose;
* Subjects who have undergone major or moderate surgery (other than for diagnosis or biopsy) within 28 days prior to the first dose, or are expected to undergo major surgery during the study;
* Subjects with severe chronic obstructive pulmonary disease (COPD) (Global Initiative for Chronic Obstructive Lung Disease [GOLD] ≥ Grade 3), or who have had intestinal adhesions or intestinal obstruction within 6 months prior to the first dose;
* Subjects with severe cardiovascular diseases, such as New York Heart Association (NYHA) Heart Disease (Class III or higher), myocardial infarction within 6 months, current unstable angina, or uncontrolled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg);
* Subjects with uncontrolled primary brain tumors or central nervous system (CNS) metastases, with significant intracranial hypertension or neuropsychiatric symptoms;
* Subjects with uncontrollable neuropsychiatric diseases, mental disorders, or substance abuse, which may affect trial compliance;
* Subjects with active infections requiring systemic treatment;
* Subjects with a known history of human immunodeficiency virus (HIV) infection;
* Subjects with hepatitis B virus (HBV) infection (HBsAg-positive or HBcAb-positive, with HBV-DNA ≥ 2000 IU/mL or HBV-DNA ≥ 10⁴ copies/mL), or hepatitis C virus (HCV) infection (HCV antibody-positive, with HCV-RNA quantitative test result above the lower limit of detection); Note: For subjects with HBV infection and HBV-DNA < 2000 IU/mL or HBV-DNA < 10⁴ copies/mL, those who are willing to receive antiviral therapy (such as entecavir, tenofovir, or other antiviral drugs) based on clinical judgment during the study may be enrolled;
* Subjects with medical history, diseases, treatments, or laboratory abnormalities that may interfere with trial results, prevent the subject from completing the entire study, or are deemed by the investigator as not being in the subject's best interest to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Adverse Events (AE); Recommended Phase 1 Clinical Dose | At the begin of Cycle 1(each cycle is 21 days)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At the end of Cycle 1(each cycle is 21 days)
Patient - reported outcome (PRO) | At the begin of Cycle 1(each cycle is 21 days)
Nutritional scale score | baseline period
  Appetite, body weight, muscle strength, vitality, serum protein levels (related to liver function), etc.

OTHER OUTCOMES:
White Blood Cell Count | At the begin and end of Cycle 1(each cycle is 21 days)
Neutrophil Count and Proportion | At the begin and end of Cycle 1(each cycle is 21 days)
Lymphocyte Count and Proportion | At the begin and end of Cycle 1(each cycle is 21 days)
Monocyte Count and Proportion | At the begin and end of Cycle 1(each cycle is 21 days)
Eosinophil Count and Proportion | At the begin and end of Cycle 1(each cycle is 21 days)
Basophil Count and Proportion | At the begin and end of Cycle 1(each cycle is 21 days)
Blood Glucose | At the begin and end of Cycle 1(each cycle is 21 days)
Triglycerides | At the begin and end of Cycle 1(each cycle is 21 days)
Safety Endpoints: Including adverse events (AEs), serious adverse events (SAEs), laboratory test abnormalities, electrocardiogram (ECG) abnormalities, and others. | On the 1st day of each 21-day treatment cycle.

IPD SHARING:
Plan to Share IPD: No